CLINICAL TRIAL: NCT01224795
Title: A Phase III, Multicenter, Randomized, Double-blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Intravenous Peramivir in Subjects With Uncomplicated Influenza.
Brief Title: A Study to Evaluate the Efficacy and Safety of Intravenous Peramivir in Subjects With Uncomplicated Influenza.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated for administrative reasons
Sponsor: BioCryst Pharmaceuticals (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCX1812-304; HHS 0100200700032C (Other Grant/Funding Number: HHS-BARDA)
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2014-12

CONDITIONS: Influenza
Keywords: uncomplicated influenza
MeSH Terms: conditions — Influenza, Human | interventions — peramivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peramivir (Experimental): Adults (≥ 18 years): Peramivir 600 mg, administered intravenously. Adolescents (12 to < 18 years): Peramivir 10 mg/kg (not to exceed a maximum dose of 600 mg), administered intravenously.
  Interventions: Drug: Peramivir
- Placebo (Placebo Comparator): Placebo Peramivir, administered intravenously.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Peramivir — Adults (≥ 18 years): Peramivir 600 mg, administered intravenously. Adolescents (12 to < 18 years): Peramivir 10 mg/kg (not to exceed a maximum dose of 600 mg), administered intravenously.
  Arms: Peramivir
Drug: Placebo Comparator — Placebo Peramivir, administered intravenously.
  Arms: Placebo

SUMMARY:
This is a study to evaluate the efficacy and safety of a single dose of intravenous peramivir versus placebo in adolescents and adults with acute uncomplicated influenza.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of a single dose of intravenous peramivir versus placebo in adolescents and adults with acute,uncomplicated influenza.

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female subjects age ≥12 years.
* Test positive for influenza A or B by Rapid Antigen Test (RAT) performed with a commercially available test on an adequate anterior nasal specimen in accordance with the manufacturer's instructions.
* Presence of at least one respiratory symptom (cough, sore throat, or nasal symptoms) of at least moderate severity.
* Presence of at least one constitutional symptom (myalgia [aches and pains], headache,feverishness, or fatigue) of at least moderate severity.
* Onset of symptoms no more than 36 hours before presentation for screening.
* Written informed consent/assent.

Exclusion Criteria:

* Women who are pregnant or breast-feeding.
* Employees of the study site, or immediate family members of study site employees.
* Presence of clinically significant signs of acute respiratory distress.
* History of severe chronic obstructive pulmonary disease (COPD) or severe persistent asthma.
* History of heart failure or angina requiring daily pharmacotherapy with symptoms consistent with New York Heart Association Class III or IV functional status within the past 12 months.
* History of chronic renal impairment requiring hemodialysis and/or known or suspected to have moderate or severe renal impairment (actual or estimated creatinine clearance <50 mL/min).
* Clinical evidence of worsening of any chronic medical condition (temporally associated with the onset of symptoms of influenza) which, in the investigator's opinion, indicates that such finding(s) could represent complications of influenza.
* Current clinical evidence, including clinical signs and/or symptoms consistent with otitis media,bronchitis, sinusitis and/or pneumonia, or active bacterial infection of any body site that requires therapy with oral or systemic antibiotics.
* Presence of immunocompromised status due to chronic illness, previous organ transplant, or use of immunosuppressive medical therapy which would include oral or systemic treatment with > 10 mg ic treatment with > 10 mg prednisone or equivalent on a daily basis within 30 days of screening.
* Presence of known HIV infection with a CD4 count <350 cell/mm3.
* Receipt of any dose of rimantadine, amantadine, zanamivir, or oseltamivir in the 7 days prior to screening.
* Immunization against influenza with live attenuated virus vaccine (FluMist®) in the previous 21 days.
* History of alcohol abuse or drug addiction within 1 year prior to admission in the study.
* Participation in a previous study of intramuscular or intravenous peramivir, or previous exposure to peramivir.
* Participation in a study of any investigational drug or device within the last 30 days.
* Presence of any pre-existing illness that, in the opinion of the investigator, would place the subject at an unreasonably increased risk through participation in this study.
* Presence of any pre-existing illness that in the opinion of the investigator would make the subject unable to comply with the protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of peramivir administered intravenously compared to placebo on the time to alleviation of clinical symptoms with acute uncomplicated influenza. | 14 Days
  Time to alleviation of clinical symptoms in adolescents and adults with uncomplicated acute influenza measured from patient reported study diaries.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of peramivir administered intravenously | 14 Days
  To evaluate time to resolution of fever in response to treatment. To evaluate changes in influenza virus titer in nasal and pharyngeal samples (viral shedding) in response to treatment.
  To evaluate secondary clinical outcomes and changes in virus susceptibility to neuraminidase inhibitors in response to treatment.

CONTACTS AND LOCATIONS:
Locations (96):
- United States (96):
  - Birmingham, Alabama
  - Hot Springs, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Mountain Home, Arkansas
  - Anaheim, California
  - Buena Park, California
  - Chino, California
  - Dinuba, California
  - Garden Grove, California
  - Lincoln, California
  - Los Angeles, California
  - Oceanside, California
  - Palm Springs, California
  - Port Hueneme, California
  - Sacramento, California
  - San Diego, California
  - Tustin, California
  - West Covina, California
  - Boulder, Colorado
  - Centennial, Colorado
  - Wheat Ridge, Colorado
  - Milford, Connecticut
  - Brooksville, Florida
  - Coral Gables, Florida
  - Cutler Bay, Florida
  - Daytona Beach, Florida
  - Edgewater, Florida
  - Gainsville, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - South Miami, Florida
  - West Palm Beach, Florida
  - Stockbridge, Georgia
  - Boise, Idaho
  - Aurora, Illinois
  - Bloomingdale, Illinois
  - Chicago, Illinois
  - Peoria, Illinois
  - South Bend, Indiana
  - Dubuque, Iowa
  - Arkansas City, Kansas
  - Lenexa, Kansas
  - Bardstown, Kentucky
  - Hazard, Kentucky
  - Paducah, Kentucky
  - Baton Rouge, Louisiana
  - Shreveport, Louisiana
  - Bangor, Maine
  - Hollywood, Maryland
  - Rockville, Maryland
  - Brockton, Massachusetts
  - Fall River, Massachusetts
  - Washington, Missouri
  - Bozeman, Montana
  - Fremont, Nebraska
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Albuquerque, New Mexico
  - Camillus, New York
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Akron, Ohio
  - Dayton, Ohio
  - Wadsworth, Ohio
  - Owasso, Oklahoma
  - Bend, Oregon
  - Medford, Oregon
  - Hatfield, Pennsylvania
  - Philadelphia, Pennsylvania
  - Scotland, Pennsylvania
  - Cranston, Rhode Island
  - Cumberland, Rhode Island
  - Johnston, Rhode Island
  - Easley, South Carolina
  - Greenville, South Carolina
  - Bristol, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - Beaumont, Texas
  - Bryan, Texas
  - Dallas, Texas
  - Forth Worth, Texas
  - Georgetown, Texas
  - Houston, Texas
  - Lake Jackson, Texas
  - North Richland Hills, Texas
  - San Antonio, Texas
  - Spring, Texas
  - Salt Lake City, Utah
  - South Jordan, Utah
  - West Jordan, Utah
  - Arlington, Virginia
  - Charlottesville, Virginia